CLINICAL TRIAL: NCT06044441
Title: ENABLE-SG (Educate, Nurture, Advise, Before Life Ends for Singapore) as a Proactive Palliative Care Model: Evaluation and Implementation Preparation
Brief Title: Evaluation and Implementation Preparation of a Proactive Palliative Care Model (ENABLE-SG)
Acronym: ENABLE-SG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ENABLE-SG; HCSAINV23jan-0001 (Other Grant/Funding Number: NMRC - HPHSR Clinician Scientist Award (HCSA))
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms
Keywords: Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENABLE-SG (immediate group) (Experimental): * Participants will receive the ENABLE-SG model immediately (six sessions for patients and four sessions for caregivers) at an approximately weekly interval.
  * Interventions: ENABLE-SG model
  Interventions: Behavioral: ENABLE-SG model
- Wait-list control (Other): * 6-month wait-list control. Participants will receive the ENABLE-SG model six months after baseline (six sessions for patients and four sessions for caregivers) at an approximately weekly interval.
  * Interventions: ENABLE-SG model
  Interventions: Other: Wait-list control

INTERVENTIONS:
Behavioral: ENABLE-SG model — Patients and caregivers will receive individual structured psycho-educational sessions with a health coach. These sessions will be primarily delivered over the phone. Patient and caregiver dyads will have different health coaches. Patients will have six sessions on the topics of maintaining positivity, self-care, coping with stress, managing symptoms, exploring what matters most, and life review. Caregivers will have four sessions on the topics of maintaining positivity, self-care, coping with stress, and managing symptoms. All sessions will begin with screening for distress using the Distress Thermometer and Problem List culturally adapted from the National Comprehensive Cancer Network. From screening results, the health coach can flexibly change the order of the topics to address specific problems. It will take approximately three months to complete all sessions.
  Arms: ENABLE-SG (immediate group)
Other: Wait-list control — * 6-month wait-list control. Participants will receive the ENABLE-SG model six months after baseline (six sessions for patients and four sessions for caregivers) at an approximately weekly interval.
  * Interventions: ENABLE-SG model
  Arms: Wait-list control

SUMMARY:
The current interdisciplinary specialist palliative care model focuses on supporting patients with advanced cancer who have complex problems in the last weeks of life. Consequently, palliative care is often provided late and in response to uncontrolled symptoms during crises. Palliative care models should shift from this reactionary illness-stress paradigm to a proactive health-wellness approach that is integrated early in the patient's disease trajectory.

A proactive early palliative care telehealth model, ENABLE (Educate, Nurture, Advise, Before Life Ends), was developed in the U.S. to coach patients with advanced cancers and their family caregivers on how to cope effectively with serious illness. By empowering individuals early before acute distress and symptoms occur, patients and families can better mitigate and avoid crises. Building on positive health outcomes demonstrated by the ENABLE model in the U.S., the study team has successfully pilot-tested a culturally adapted ENABLE-SG model in Singapore. This study seeks to test the effectiveness of this ENABLE-SG model among patients with recently diagnosed advanced cancer and their caregivers while simultaneously collecting data on real-world implementation.

DETAILED DESCRIPTION:
To evaluate the effectiveness of the ENABLE-SG model, we will conduct a randomized wait-list controlled trial comparing clinical outcomes at 6 months between patients and caregivers receiving early ENABLE-SG and their wait-listed counterparts receiving usual care. Eligible patients and their caregivers will be randomly assigned at baseline to receive ENABLE-SG either immediately or after a 6-month waiting period. To evaluate ways to improve implementation, the Consolidated Framework for Implementation Research (CFIR) will be used to systematically identify processes that influence implementation outcomes.

The specific aims and hypotheses of this study are:

1. Assess the effectiveness of ENABLE-SG among patients with advanced cancer. We hypothesize that at 6 months, compared to usual care, patients who received ENABLE-SG will have better health-related quality of life (QoL), mood, health status, coping strategies, lesser palliative care concerns, lesser acute healthcare utilisation, and smaller hospital bill size. At 12 months, compared to wait-list control group, early ENABLE-SG recipients will have better primary and secondary outcomes.
2. Assess the effectiveness of ENABLE-SG among caregivers of patients with advanced cancer. We hypothesize that at 6 months, compared to usual care, caregivers who received ENABLE-SG will have better caregiver health-related QoL, mood, coping strategies, satisfaction with care, and lower caregiving costs. At 12 months, compared to wait-list control group, early ENABLE-SG recipients will have better primary and secondary outcomes.
3. Assess ways to improve ENABLE-SG implementation in the real-world context.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients:

  1. Adult aged 21 and above
  2. Within 60 days of being informed of an advanced cancer diagnosis, defined as metastatic or recurrent/ progressive Stage III/IV solid tumour
  3. Able to speak English or Chinese
  4. Able to provide informed consent
  5. Patients will NOT need to have a caregiver willing to participate in the ENABLE-SG programme.
* Inclusion criteria for caregivers:

  1. Adult aged 21 and above
  2. Self-endorsing or identified by the enrolled patient as an unpaid spouse/partner, relative or friend who knows them well and who provides regular support (at least 7 hours a week) due to their cancer and who does not have to live in the same dwelling
  3. Caring for a patient with advanced cancer (see definition under patient inclusion criteria above)
  4. Able to speak English or Chinese.
  5. Able to provide informed consent
* Inclusion criteria for healthcare professions:

  1. 21 years or older.
  2. Approached to participate in the ENABLE-SG study
  3. Able to provide informed consent

Exclusion Criteria:

* Exclusion criteria for patients:

  1. Medical record documentation of an active severe mental illness, dementia, active suicidal ideation, uncorrected hearing loss
  2. Unable to complete patient-reported outcome measures
  3. Has been reviewed by palliative care services in the current model of palliative care.
* Exclusion criteria for caregivers:

  1. Self-reported severe mental illness, dementia, active suicidal ideation, uncorrected hearing loss
  2. Unable to complete caregiver-reported outcomes.
* Exclusion criteria for healthcare professional:

  1. Healthcare professionals that are not providing care for cancer patients.
  2. Unable to complete interviews.

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 715 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life of patients with advanced cancer | 6th month.
  Quality of life score measured using the Functional Assessment of Chronic Illness Therapy - Palliative (FACIT-Pal), a 46-item measure with a quality of life scale (4 domains: physical, emotional, social, and functional well-being) and a palliative care subscale. It has demonstrated internal consistency, reliability and validity for persons with advanced cancer. Scores range from 0 to 184, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Health-related quality of life of caregivers | 6th month.
  Quality of life score measured using the Singapore Caregiver Quality of Life Scale (SCQOLS), a 15-item quality of life measure covering 5 domains: physical well-being, mental well-being, experience & meaning, impact on daily living, and financial well-being. The domain scores will be scaled to range from 0 to 100, with a higher score indicating better quality of life.
Longitudinal changes in health-related quality of life of patients with advanced cancer across assessment timepoints | Baseline, 3rd month, 6th month, 9th month, 12th month.
  Longitudinal changes in quality of life score measured using the Functional Assessment of Chronic Illness Therapy - Palliative (FACIT-Pal), across assessment timepoints. FACIT-Pal is a 46-item measure with a quality of life scale (4 domains: physical, emotional, social, and functional well-being) and a palliative care subscale. It has demonstrated internal consistency, reliability and validity for persons with advanced cancer. Scores range from 0 to 184, with higher scores indicating better quality of life.
Longitudinal changes in health-related quality of life of caregivers across assessment timepoints | Baseline, 3rd month, 6th month, 9th month, 12th month.
  Longitudinal changes in quality of life score measured using the Singapore Caregiver Quality of Life Scale (SCQOLS), across assessment timepoints. SCQOLS is a 15-item quality of life measure covering 5 domains: physical well-being, mental well-being, experience & meaning, impact on daily living, and financial well-being. The domain scores will be scaled to range from 0 to 100, with a higher score indicating better quality of life.
Mood of patients with advanced cancer and their caregivers | Baseline, 3rd month, 6th month, 9th month, 12th month.
  Mood measured using the Center for Epidemiological Studies-Depression (CES-D), a 20-item measure of symptoms clustered in 4 domains: depressed affect, somatic complaints, positive affect, and interpersonal activity. Scores will be scored to a total score ranging from 0 to 60, with higher scores indicating greater frequency of depressive experiences.
Coping strategies of patients with advanced cancer and their caregivers | Baseline, 3rd month, 6th month, 9th month, 12th month.
  Coping strategies measured using the Brief Coping Orientation to Problems Experienced (Brief-COPE) Inventory, a 28-item measure of coping strategies in 14 subscales: self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, behavioural disengagement, venting, positive reframing, planning, humour, acceptance, religion, and self-blame. This scale has been validated in the cancer population. Each subscale score will be derived from the sum of two corresponding items scored on a 4-point Likert scale from "I do not do this at all" to "I usually do this a lot".
Palliative care concerns of patients with advanced cancer | Baseline, 3rd month, 6th month, 9th month, 12th month.
  Palliative care concerns measured using the Integrated Palliative Care Outcomes Scale (IPOS), a brief measure of palliative care problems, covering physical and psychological symptoms, social and spiritual issues, communication, information needs, and practical concerns. The scores on all items will be summed to give a total score ranging from 0 to 40, with higher scores indicating more care needs.
Health states of patients with advanced cancer | Baseline, every 3 months until death or end of the study.
  Health states measured using the EuroQOL Group 5-Dimension Health-related Quality of Life Measurement (EQ-5D-5L), which contains a 5-item descriptive system measuring 5 dimensions: mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression; a visual analogue scale measuring overall health status.
Healthcare resource utilization of patients with advanced cancer | Baseline until death or end of the study.
  The following data will be extracted from electronic medical records: dates of emergency department visits and hospital admissions, hospital bill size, date of first review by existing palliative care services, date of death, and place of death.
Caregivers' satisfaction with care | Baseline, 3rd month, 6th month, 9th month, 12th month.
  Satisfaction with care measured using the Family Satisfaction with End-of-Life Care (FAMCARE) Scale, a 10-item unidimensional scale measuring family satisfaction. Scores on all items will be summed to give a total score ranging from 0 to 20, with higher scores indicating higher satisfaction levels.
Healthcare resource utilization of caregivers | Baseline, 3rd month, 6th month, 9th month, 12th month.
  Healthcare resource utilization and caregiving cost. A questionnaire recording employment status and productivity loss (hours missed from work, impairment while at work, and impairment in regular activities) due to caregiving. The following data will be extracted from electronic medical records: dates of emergency department visits and hospital admissions, and hospital bill size.

OTHER OUTCOMES:
Acceptability and adoption of ENABLE-SG among patients with advanced cancer and their caregivers. | At the end of study participation, up to the 12th month.
  An investigator-designed structured feedback survey on acceptability, relevance, comfort level, overall satisfaction, and intention to recommend ENABLE-SG to others in similar situations. All items are rated on a 5-point Likert scale.
Appropriateness and feasibility of ENABLE-SG among patients with advanced cancer, their caregivers, and healthcare providers | ≥6 months after baseline.
  Semi-structured interviews conducted using an interview guide developed based on the Consolidated Framework for Implementation Research (CFIR).
Fidelity of the delivery of ENABLE-SG | Through study completion, anticipated up to 3 years.
  Fidelity to the health coaching protocol (intervention) will be assessed by a narrative synthesis of any modifications or deviations from the protocol. These modifications/ deviations will be extracted from self-reporting checklists, field notes, recordings of the actual health coaching sessions, and discussions of the completed health coaching sessions.
Implementation cost | Through study completion, anticipated up to 3 years.
  Process maps and project records detailing key intervention activities to elucidate cost of involved personnel and resources through a time-tracking system and an activity-based costing approach.
Penetration | Through study completion, an average of 2 years.
  Based on study records, the Number and proportion of approached oncologists who agree for study to be conducted in their clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Grace M Yang, MRCP, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hui D, Bruera E. Models of Palliative Care Delivery for Patients With Cancer. J Clin Oncol. 2020 Mar 20;38(9):852-865. doi: 10.1200/JCO.18.02123. Epub 2020 Feb 5. PMID 32023157
- [Background] Bakitas M, Stevens M, Ahles T, Kirn M, Skalla K, Kane N, Greenberg ER; Project Enable Co-Investigators. Project ENABLE: a palliative care demonstration project for advanced cancer patients in three settings. J Palliat Med. 2004 Apr;7(2):363-72. doi: 10.1089/109662104773709530. PMID 15130218
- [Background] Maloney C, Lyons KD, Li Z, Hegel M, Ahles TA, Bakitas M. Patient perspectives on participation in the ENABLE II randomized controlled trial of a concurrent oncology palliative care intervention: benefits and burdens. Palliat Med. 2013 Apr;27(4):375-83. doi: 10.1177/0269216312445188. Epub 2012 May 9. PMID 22573470
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Background] Bakitas MA, Tosteson TD, Li Z, Lyons KD, Hull JG, Li Z, Dionne-Odom JN, Frost J, Dragnev KH, Hegel MT, Azuero A, Ahles TA. Early Versus Delayed Initiation of Concurrent Palliative Oncology Care: Patient Outcomes in the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1438-45. doi: 10.1200/JCO.2014.58.6362. Epub 2015 Mar 23. PMID 25800768
- [Background] Dionne-Odom JN, Azuero A, Lyons KD, Hull JG, Tosteson T, Li Z, Li Z, Frost J, Dragnev KH, Akyar I, Hegel MT, Bakitas MA. Benefits of Early Versus Delayed Palliative Care to Informal Family Caregivers of Patients With Advanced Cancer: Outcomes From the ENABLE III Randomized Controlled Trial. J Clin Oncol. 2015 May 1;33(13):1446-52. doi: 10.1200/JCO.2014.58.7824. Epub 2015 Mar 23. PMID 25800762
- [Derived] Ke Y, Cheung YB, Bakitas M, Odom JN, Lum E, Tan DSW, Tan TJ, Finkelstein E, Oh HC, Zhou S, Yang GM. ENABLE-SG (Educate, Nurture, Advise, Before Life Ends for Singapore) as a proactive palliative care model: protocol for a hybrid type 1 effectiveness-implementation randomized wait-list controlled trial. BMC Palliat Care. 2024 Jan 30;23(1):29. doi: 10.1186/s12904-024-01353-2. PMID 38287335